CLINICAL TRIAL: NCT01637259
Title: Maraviroc Switch Collaborative Study Renal Substudy
Brief Title: MARCH Renal Substudy
Acronym: MARCHrenal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: MARCH-Kirby renal
Record Dates: First submitted 2012-06-27; First posted 2012-07-11 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Proteinuria; HIV
Keywords: proteinuria; HIV
MeSH Terms: conditions — Proteinuria | interventions — Tenofovir; Emtricitabine; Zidovudine; abacavir; Lamivudine; Atazanavir Sulfate; Lopinavir; Darunavir; fosamprenavir; Ritonavir; Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NRTI + PI (Active Comparator): arm 1
  Interventions: Drug: arm 1 nucleotide analogue reverse transcriptase inhibitors and boosted protease inhibitors
- PI + maraviroc (Active Comparator): arm 2
  Interventions: Drug: Arm 2 boosted protease inhibitors and maraviroc
- NRTI + maraviroc (Active Comparator): arm 3
  Interventions: Drug: Arm 3 nucleotide analogue reverse transcriptase inhibitors and maraviroc

INTERVENTIONS:
Drug: arm 1 nucleotide analogue reverse transcriptase inhibitors and boosted protease inhibitors — NRTI + PI
  Other Names: tenofovir; emtricitabine; zidovudine; abacavir; lamivudine; atazanavir; lopinavir; darunavir; fosamprenavir; ritonavir
  Arms: NRTI + PI
Drug: Arm 2 boosted protease inhibitors and maraviroc — PI + maraviroc
  Other Names: maraviroc; atazanavir; lopinavir; darunavir; fosamprenavir; ritonavir
  Arms: PI + maraviroc
Drug: Arm 3 nucleotide analogue reverse transcriptase inhibitors and maraviroc — NRTI + maraviroc
  Other Names: maraviroc; tenofovir; emtricitabine; zidovudine; abacavir; lamivudine
  Arms: NRTI + maraviroc

SUMMARY:
Chronic kidney disease (CKD) is an emerging problem in patients with treated HIV. Antiretroviral therapy associated renal dysfunction has been predominantly described in terms of reduced glomerular filtration (eGFR). Proteinuria is a key component of CKD and may occur in the absence of significant reductions in eGFR. This substudy is an exploration of changes in urinary protein excretion in a randomised, open-label study to evaluate the efficacy and safety of MVC as a switch for either nucleoside or nucleotide analogue reverse transcriptase inhibitors (N(t)RTI) or boosted protease inhibitors (PI/r) in HIV-1 infected individuals with stable, well-controlled plasma HIV-RNA while taking their first N(t)RTI + PI/r regimen of combination antiretroviral therapy (cART).

DETAILED DESCRIPTION:
The aim of this substudy of MARCH is to characterize the changes in protein and salt excretion through the kidney utilising the randomised arms of the parent study MARCH. The investigators hypothesize there will be an improvement in proteinuria in those switching to maraviroc containing regimens.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written, informed consent for participation in the substudy
* Enrolled into the substudy either at or before the week 0 visit of the main study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
changes in proteinuria and albuminuria between baseline and week 96 | 96 weeks
  To compare the change in protein and albumin excretion as measured by the urine PCR and ACR through the kidneys between the randomised and standard of care (control) arm of MARCH.

SECONDARY OUTCOMES:
changes in renal tubular function between baseline and week 96 | 96 weeks
  To evaluate the following aspects of renal function at baseline and changes within and between study groups:
  * Tubular function defined as proximal tubular function; ascending thick loop of Henle; distal tubular function; volume and renal potassium handling;
  * Non-tubular function i.e. eGFR; Urine albumin:creatinine ratio;
  * Determine factors associated with renal dysfunction within the cohort e.g. demographics, HIV related, HIV-treatment related, co-morbidities, concomitant medication (such as ACE inhibitors and ARB; PI/r co-administered with TDF); TDF use;

CONTACTS AND LOCATIONS:
Overall Officials: Waldo Belloso, MD, Principal Investigator — Hospital Italiano de Buenos Aires; Mark Kelly, MD, Principal Investigator — Brisbane Sexual Health and HIV Service
Locations (15):
- Argentina (3):
  - Hospital Italiano de Buenos Aires, Buenos Aires, Buenos Aires F.D.
  - Hospital General de Agudos J M Ramos Mejia, Buenos Aires, Buenos Aires F.D.
  - Fundación IDEAA, Buenos Aires, Buenos Aires F.D.
- Australia (2):
  - St. Vincent's Hospital, Sydney, New South Wales
  - Brisbane Sexual Health and HIV Service, Brisbane, Queensland
- Canada (3):
  - Southern Alberta Clinic, Calgary, Alberta
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - Clinic Opus/Lori, Montreal, Quebec
- Germany (2):
  - Klinikum der Universitat Zu Koln, Cologne
  - Universitätsklinikum Düsseldorf, Klinik für Gastroenterologie, Hepatologie und Infektiologie, MX-Ambulanz, Düsseldorf
- Nagoya Medical Center, Nagoya, Japan
- Instituto Nacional de Ciencias Medicas y Nutriciòn Salvador Zubiran, Mexico City, Tlalpan DF, Mexico
- Chulalongkorn University Hospital, Bangkok, Thailand
- United Kingdom (2):
  - Western General Hospital, Edinburgh, Lothian
  - Brighton & Sussex University NHS Trust, Brighton, Sussex